CLINICAL TRIAL: NCT00184392
Title: Debridement After Functional Endoscopic Sinus Surgery
Brief Title: Cleaning of the Nose After Sinus Surgery: Necessary or Only Bothersome?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Midt-Norge (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 229-04
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Acute Recurrent Rhinosinusitis
Keywords: Sinus surgery; endoscopic; postoperative care; debridement; randomized; acute recurrent rhinosinusitis; chronic rhinosinusitis; nasal polyps; Chronic rhinosinusitis with nasal polyps; Chronic rhinosinusitis without nasal polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Debridement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- debridement or saline irrigation (Experimental): 1 arm undergo debridement of the nose 1 week and 2 weeks after surgery the other arm rinse their nose with saline irrigation
  Interventions: Procedure: debridement or saline irrigation

INTERVENTIONS:
Procedure: debridement or saline irrigation — debridement of crusts, blood and secretions from the nose 1 week and 2 weeks after surgery

SUMMARY:
The goal of this study is to increase knowledge about how to treat patients after sinus surgery.

DETAILED DESCRIPTION:
Many surgeons consider the postoperative treatment after sinus surgery as important for the outcome as the surgery itself. However, postoperative treatment regimes differ considerably between surgeons. They include non-intervention, frequent in-office endoscopic debridement, stenting of the middle meatus, saline douching or irrigation of the nose, or combinations of these measures in various ways. The lack of consensus is unfortunate. It indicates a lack of knowledge about how to treat these patients optimally after surgery. This is partly due to a lack of internationally acknowledged randomised, comparative, prospective studies on the effects of the various postoperative measures and their interactions. Accordingly, some patients may receive a too intensive postoperative follow up, with unnecessary frequent visits with the doctor, unnecessary bleeding and inconvenience from unnecessary debridement/cleaning of the nose, and increased costs due to unnecessary medication. Conversely, there may be patients that receive too little attention in the postoperative period, and thus may have a suboptimal result of the operation.

Frequent cleaning/debridement of the nose after sinus surgery is believed to improve the outcome of functional endoscopic sinus surgery (FESS). However, the scientific data on its effects are limited. The purpose of this study was to evaluate the effects of cleaning/ debridement of the middle meatus 5-7 days and 12-14 days after sinus surgery in a randomized, partly blinded, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria are acute recurrent rhinosinusitis and chronic rhinosinusitis. The investigators used the classification of rhinosinusitis proposed by Lanza and Kennedy.

Exclusion Criteria:

* Previous FESS
* Systemic disease with affection of the nose (Wegener's granulomatosis, cystic fibrosis, Kartagener's syndrome, sarcoid)
* Primary ciliary dyskinesia
* Pregnancy
* Septoplasty in the same surgery
* Ongoing treatment for cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Primary Completion 2005-12 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Adhesions in middle meatus or not | 3 months
  synechia between concha media and lateral nasal wall 0=no adhesion
  1=adhesions present

SECONDARY OUTCOMES:
Pain due to cleaning of the nose | 1 and 2 weeks after surgery
  Pain on VAS
Does cleaning of the nose reduce: crusts in the nose 14 days after surgery | 2 weeks after surgery
  0=no crusts
  1. =mild
  2. =impossible to see under concha media
the tendency to post operative infections | 3 months
  Patient information connected to examination from the investigator
Does debridement increase bleeding from the nose the first 14 days after surgery | 2 weeks
  0 no bleeding
  1. spots of blood
  2. bleeding from the nose
nasal congestion after surgery | 2 weeks
  a patient diary, the patient mark nasal congestion on a VAS from day 1 to day 14 after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Bugten, M.D., Principal Investigator — Department of Otolaryngology, Head and Neck Surgery, St Olav University Hospital of Trondheim, and Norwegian University of Science and Technology (NTNU), 7006 Trondheim, Norway
Locations (2):
- Norway (2):
  - Department of Otolaryngology, Sorlandet Hospital, Kristiansand
  - Department of Otolaryngology, Head and Neck Surgery, St Olav University Hospital of Trondheim, and Norwegian University of Science and Technology (NTNU), 7006 Trondheim, Norway, Trondheim

REFERENCES:
- [Result] Bugten V, Nordgard S, Steinsvag S. The effects of debridement after endoscopic sinus surgery. Laryngoscope. 2006 Nov;116(11):2037-43. doi: 10.1097/01.mlg.0000241362.06072.83. PMID 17075402